CLINICAL TRIAL: NCT00189631
Title: UFT/LV Maintenance Vs Observation in Metastatic Breast Cancer Responsive to Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Européenne de Recherche en Oncologie (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AERO-MB02
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-12-08 (Estimated); Status verified 2005-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

INTERVENTIONS:
Procedure: UFT/LV
Procedure: Observation

SUMMARY:
To compare maintenance therapy to observation in metastatic breast cancer patients responding (or stabilized) after 1st-line chemotherapy. Main endpoint is disease-free survival. Secondary endpoints are overall survival and tolerance. A total of 200 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* metastatic breast cancer
* objective response or stabilisation after 6 to 8 cycle of a first line chemotherapy
* time period between the end of chemotherapy and randomization < 4 weeks
* age over 18 years
* Performance status (OMS) < 2.
* Life expectancy > 3 months
* Biological criteria before randomization: Neutrophiles > 1.5 x 109 G/L; Pl. > 100 x 109 G/L; Hb > 10 g/dl; Creatininemia < 1,5 UNL; Bili. < 2 UNL; Transaminases < 2,5 UNL; Alcalines Phosphatases < 2,5 UNL
* Signed written informed consent

Exclusion Criteria:

* Metastatic breast cancer having received more than one chemotherapy line.
* Tumor progression under chemotherapy
* Free interval between primary tumor and metastases > 5 years, with estrogen receptors and without visceral metastases
* Free interval between primary tumor and metastases < 18 months after adjuvant chemotherapy if first lime chemotherapy only led to a tumor stabilization
* Concomitant hormonotherapy
* Other cancer
* Symptomatic brain metastases
* Any uncontrolled severe disease except breast cancer (especially cardiac failure with LVEF < 50% or coronary insufficiency
* Psychiatric disorder
* Other concomitant trial
* Male patient
* Pregnancy and breast-feeding (effective contraception is mandatory in the case of women of child-bearing potential)
* History of high dose chemotherapy with bone marrow transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Berdah, MD, Principal Investigator — AERO; Laurent Zelek, MD, Principal Investigator — AERO; Bruno Audhuy, MD, Principal Investigator — AERO
Locations (1):
- AERO, Créteil, France